CLINICAL TRIAL: NCT07068776
Title: Shockwave Intervention for Enhanced Wound Healing in No-touch Pedicle Saphenous Vein Graft Harvesting for Coronary Artery Bypass Grafting: A Prospective, Single-Center, Single-Blind, Randomized, Sham-Controlled Study
Brief Title: Shockwave Intervention for Enhanced Wound Healing in No-touch Pedicle Saphenous Vein Graft Harvesting for Coronary Artery Bypass Grafting
Acronym: SHIELDS-CABG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1054/2025
Record Dates: First submitted 2025-06-05; First posted 2025-07-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-05

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: Coronary artery bypass grafting; Saphenous vein graft (SVG); No-touch vein harvesting; Wound healing complications; Shockwave therapy (SWT); Cardiac surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Participants in this arm receive intraoperative shockwave therapy (SWT) applied to the leg wound after saphenous vein harvesting and wound closure. Shockwaves are administered during the reperfusion phase while the patient is still on cardiopulmonary bypass. The applicator is moved in circular motion over the wound using a sterile cover and ultrasound gel. The energy settings are 0.1 mJ/mm² at 5 Hz, with 25 impulses per centimeter of wound length. This intervention aims to reduce postoperative wound healing complications.
  Interventions: Device: Shockwave treatment
- Sham group (Sham Comparator): Participants in this arm receive a sham treatment mimicking the active shockwave therapy. The applicator is moved over the leg wound in the same sterile manner using ultrasound gel and sterile cover, but no shockwaves are emitted. The procedure takes the same amount of time and follows the same protocol.
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Shockwave treatment — The shockwave device will be set to an energy flux density of 0.1 mJ/mm² at 5 Hz, with approximately 25 impulses per centimeter of wound length. This means that one centimeter of the wound will be treated for 5 seconds. The shockwave treatment will then be carried out, with each centimeter of the wound area treated for 5 seconds using gentle circular motions.
  Arms: Treatment group
Device: Sham treatment — The applicator will not be connected to the shockwave device. The applicator treatment will then be carried out, with each centimeter of the wound area treated for 5 seconds using gentle circular motions.
  Arms: Sham group

SUMMARY:
The aim of this trial is to apply shockwaves to the leg wound after saphenous vein harvesting and closure in order to reduce the occurrence of postoperative wound healing complications following coronary artery bypass grafting using venous grafts.

DETAILED DESCRIPTION:
Selection of suitable grafts for coronary artery bypass grafting (CABG) is one of the most critical decisions cardiac surgeons must make. There are two main techniques for harvesting graft vessels. The first is the skeletonized harvesting technique (ST), in which only the vessel itself is dissected and isolated before removal. The second method is the "no-touch" technique (NT), where the vessel is harvested along with surrounding tissue to minimize direct manipulation and potential microtrauma to the graft.

Saphenous vein grafts (SVG) are the most commonly used conduits in CABG and can be harvested using either technique. While the NT technique has demonstrated superior long-term patency and reduced atherosclerotic changes, it is associated with a significantly higher rate of wound healing complications, which are often more severe and can have a considerable impact on patient quality of life.

Shockwave therapy (SWT) has been shown to accelerate wound healing. The SHIELDS-CABG trial employs a double-blinded, sham-controlled design to evaluate the efficacy of prophylactic SWT in reducing wound healing complications after NT saphenous vein harvesting in CABG patients. In this study, the intervention group receives SWT immediately after wound closure to enhance healing and prevent complications.

This is a prospective, single-center, single-blinded, randomized, sham-controlled trial conducted at the Department of Cardiac Surgery, Medical University of Innsbruck. Blinding is maintained intraoperatively and only applied after wound closure to avoid procedural bias. Half of the patients will receive SWT, while in the control group the device will be held over the wound for the same duration without delivering shockwaves. A double-blind design is not feasible, as the operating staff can hear the characteristic sound of the device during SWT application.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years
* Isolated CABG procedure in the need of 2 or more venous grafts
* Elective or urgent cases
* Median sternotomy approach
* eGFR ≥ 15 ml/min
* Willing to participate in trial
* Able to provide informed consent

Exclusion Criteria:

* History of venous stripping or ligation
* Uncontrolled Diabetes mellitus (HbA1c ≥ 9 %)
* Enrolled in other therapeutic or interventional trial
* Hemodynamically unstable
* Cardiogenic shock
* Any condition that seriously increases the risk of noncompliance or loss of follow-up
* Emergency case
* Salvage case

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Wound Healing Disturbance | 30 days after surgery
  We defined the occurrence of a wound healing complication as followed:
  Definition of Surgical Site Infection (SSI)
  The SSI definition is in accordance with the guidelines of the center for disease control and their recommendations for superficial incisional SSI:
  * Date of event occurs within 30 days following the operative procedure AND involves only skin and subcutaneous tissue of the incision AND
  * Patient has at least one of the following:
    * Purulent drainage from the superficial incision
    * Organism(s) identified from an aseptically-obtained specimen from the superficial incision or subcutaneous tissue by a culture or non-culture based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment
    * Superficial incision that is deliberately opened by a sur

SECONDARY OUTCOMES:
Bates-Jensen Wound Assessment Tool | From randomization to the end of participation at 180 days
  Difference in the Bates-Jensen Wound Assessment Tool (BWAT) score. The BWAT is a validated instrument used to assess wound healing, consisting of 13 scored items related to wound size, depth, edges, undermining, necrotic tissue, exudate, skin color, peripheral tissue, granulation, and epithelialization. Each item is scored from 1 (best) to 5 (worst). The total score ranges from 13 (completely healed wound) to 65 (most severe wound condition). Higher scores indicate worse wound status.
Change in EQ-5D-5L Index Score | From randomization to end of study participation at 180 days
  Difference in the EQ-5D-5L index score, a standardized measure of health-related quality of life developed by the EuroQol Group. The EQ-5D-5L index score ranges from -0.594 to 1.000, where higher scores indicate better health status. A score of 1 represents full health, 0 represents a health state equivalent to death, and negative values represent health states considered worse than death.
Unscheduled visits | From randomization to end of study participation at 180 days
  Number of unscheduled outpatient visits
Surgical revision | From randomization to end of study participation at 180 days
  Rate of surgical revisions due to wound healing complications, except for bleeding
Antibiotics due to wound healing | From randomization to end of study participation at 180 days
  Proportion of patients requiring antibiotics due to wound healing complications
Discharge wound state | From randomization to discharge (Day 8±3)
  Wound status at discharge Difference in the Bates-Jensen Wound Assessment Tool (BWAT) score. The BWAT is a validated instrument used to assess wound healing, consisting of 13 scored items related to wound size, depth, edges, undermining, necrotic tissue, exudate, skin color, peripheral tissue, granulation, and epithelialization. Each item is scored from 1 (best) to 5 (worst). The total score ranges from 13 (completely healed wound) to 65 (most severe wound condition). Higher scores indicate worse wound status.
Laboratory values | From randomization to end of study participation at 180 days
  Difference in laboratory values:
  * HbA1c
  * Creatinin
  * Total Cholesterol
  * LDL-C
  * HDL-C
  * Lp(a)
  * LDH,
  * Erythrocytes,
  * Haemoglobin
  * Haematocrit
  * Platelet count
  * Leukocytes
  * CRP,
  * APTT,
  * INR
  * NT-pro-BNP
  * Total CK
  * CK-MB
  * CK-MB %
  * Troponin T
Adverse events | From randomization to end of study participation at 180 days
  Device related adverse events A clinical trial adverse event is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in a patient or clinical trial subject C or not related to the investigational medical device. This includes events related or not to a comparator and procedures involved.
  Surgical procedures themselves are not AEs; they are therapeutic measures for conditions that require surgery. The condition for which the surgery is required may be an AE. Planned surgical measures permitted by the clinical trial protocol and the condition(s) leading to these measures are not AEs, if the condition leading to the measure was present prior to inclusion into the trial.
Serious Adverse Events | From randomization to end of study participation at 180 days
  Device related Serious Adverse Events
  * death (excluding death from progressive disease)
  * a life-threatening experience - refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe
  * initial hospitalization, or prolongation of existing inpatients hospitalization
  * persistent or significant disability or incapacity
  * congenital anomaly or birth defect
  * occur a malignant tumor

CONTACTS AND LOCATIONS:
Overall Officials: Can Gollmann-Tepeköylü, MD, PhD, Principal Investigator — Department of Cardiac Surgery, Medical Univesity Innsbruck, Innsbruck, Austria
Locations (1):
- Department of Cardiac Surgery, Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly shared but may be made available upon reasonable request to the principal investigator.